CLINICAL TRIAL: NCT01920932
Title: Adcetris (Brentuximab Vedotin), Substituting Vincristine in the OEPA/COPDac Regimen [Treatment Group 3 (TG3) of Euro-Net C1] With Involved Node Radiation Therapy for High Risk Pediatric Hodgkin Lymphoma (HL)
Brief Title: Adcetris (Brentuximab Vedotin), Combination Chemotherapy, and Radiation Therapy in Treating Younger Patients With Stage IIB, IIIB and IV Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLHR13; NCI-2013-01123 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2013-08-06; First posted 2013-08-12 (Estimated); Results first posted 2022-02-08 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Stage II Childhood Hodgkin Lymphoma; Stage III Childhood Hodgkin Lymphoma; Stage IV Childhood Hodgkin Lymphoma
Keywords: Pediatric cancer; Hodgkin lymphoma; Targeted therapy; Frontline therapy; Brentuximab vedotin; Quality of Life; OEPA/COPDac
MeSH Terms: conditions — Neoplasms; Hodgkin Disease | interventions — Brentuximab Vedotin; Etoposide; Prednisone; Prednisolone; Doxorubicin; Cyclophosphamide; Dacarbazine; Filgrastim; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Participants receive AEPA regimen (brentuximab vedotin, etoposide, prednisone, doxorubicin), and CAPDac regimen (cyclophosphamide, brentuximab vedotin, prednisone, dacarbazine(R)). Filgrastim may be given as clinically indicated. For those with lymph nodes that do not go into remission after 2 courses of AEPA chemotherapy, radiation therapy will be given. Some participants may volunteer to complete the quality of life assessment.
  Interventions: Drug: brentuximab vedotin; Drug: etoposide; Drug: prednisone; Drug: doxorubicin; Drug: cyclophosphamide; Drug: Dacarbazine(R); Drug: filgrastim; Other: quality of life assessment; Radiation: radiation therapy

INTERVENTIONS:
Drug: brentuximab vedotin — Given intravenously (IV).
  Other Names: SGN-35; Adcetris(R)
Drug: etoposide — Given IV.
  Other Names: VP-16; Vepesid(R)
Drug: prednisone — Given orally (PO).
  Other Names: prednisolone
Drug: doxorubicin — Given IV.
  Other Names: Adriamycin(R)
Drug: cyclophosphamide — Given IV.
  Other Names: Cytoxan(R)
Drug: Dacarbazine(R) — Given IV.
  Other Names: Dimethyl Triazeno Imidazole Carboximide (DTIC)
Drug: filgrastim — Given subcutaneously (SQ) as clinically indicated.
  Other Names: Neupogen(R)
Other: quality of life assessment — Quality of life assessment will be done at initial clinical visit, and during chemotherapy, completion of therapy, then at 1 year, 2 years and 5 years. It should take no more than 15-20 minutes to complete. Participation is voluntary by participating institution and by participant.
Radiation: radiation therapy — At the end of chemotherapy and recovery of blood counts, radiotherapy will be given to any involved nodes (if any) that are not in complete remission.
  Other Names: irradiation; radiotherapy; radiation

SUMMARY:
This pilot phase II trial studies how well giving brentuximab vedotin, combination chemotherapy, and radiation therapy works in treating younger patients with stage IIB, IIIB or IV Hodgkin lymphoma. Monoclonal antibodies, such as brentuximab vedotin, can block cancer growth in different ways. Some block the ability of cancer to grow and spread. Others find cancer cells and help kill them or carry cancer killing substances to them. Drugs used in chemotherapy, such as etoposide, prednisone, doxorubicin hydrochloride, cyclophosphamide, and dacarbazine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill cancer cells. Giving brentuximab vedotin with combination chemotherapy may kill more cancer cells and reduce the need for radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* To evaluate the safety of brentuximab vedotin, etoposide, prednisone and doxorubicin hydrochloride (AEPA)/cyclophosphamide, brentuximab vedotin, prednisone and dacarbazine (CAPDac), as well as the efficacy (early complete response) after 2 cycles of AEPA chemotherapy in high risk patients with Hodgkin lymphoma (HL).
* To compare the event-free survival in high risk HL patients treated with AEPA/CAPDac to the historical control unfavorable risk 2 arm (UR2) of the St. Jude HOD99 study.

SECONDARY OBJECTIVES:

* To estimate the number of patients with adequate response according to the definitions in the Euro-Net C1 after 2 cycles of AEPA.
* To evaluate the safety of Adcetris (brentuximab vedotin) in the AEPA/CAPDac regimen in children with high risk HL.
* To describe acute hematologic, neuropathic, and infectious toxicities as they relate to transfusion requirements, growth factor support, episodes of febrile neutropenia and hospitalizations, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0.
* To study the association between local failure and original lymph node region and volume of radiation (patterns of treatment failure).
* To assess patient-reported symptoms and health-related quality of life in children with high risk HL compared to those treated on the unfavorable treatment arm of the St. Jude HOD99 study.

OUTLINE:

AEPA REGIMEN: Patients receive brentuximab vedotin on days 1, 8, and 15, etoposide on days 1 to 5, prednisone three times daily (TID) on days 1 to 15, and doxorubicin hydrochloride on days 1 and 15. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity.

CAPDac REGIMEN: Patients receive cyclophosphamide on days 1 and 8, brentuximab vedotin days 1 and 8, prednisone TID on days 1 to 15, and dacarbazine on days 1 to 3. Treatment repeats every 21-28 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Beginning 2-3 weeks after CAPDac chemotherapy, patients with lymph nodes that do not go into remission after 2 courses of AEPA chemotherapy undergo radiation therapy daily, 5 days a week for 3-4 weeks.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 4 months for 2 years, every 6 months for 2 years, and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, previously untreated CD30+ classical Hodgkin Lymphoma (HL). (Participants receiving limited emergent radiation therapy (RT) or steroid therapy - maximum of 7 days - because of cardiopulmonary decompensation or spinal cord compression will be eligible for protocol enrollment).
* Age ≤ 18 years at the time of diagnosis (i.e., participants are eligible until their 19th birthday).
* Ann Arbor stage IIB, IIIB, IVA, or IVB.
* Adequate renal function based on GFR ≥ 70 ml/min/1.73m^2 or serum creatinine adjusted for age and gender.
* Adequate hepatic function (total bilirubin < 1.5 x ULN for age, and SGOT/SGPT < 2.5 x ULN for age).
* Female participant who is post-menarchal must have a negative urine or serum pregnancy test.
* Female or male participant of reproductive potential must agree to use an effective contraceptive method throughout duration of study treatment.

Exclusion Criteria:

* CD30 negative HL.
* Has received prior therapy for Hodgkin lymphoma, except as noted above.
* Inadequate organ function as described above.
* Inability or unwillingness of research participant or legal guardian / representative to give written informed consent.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 77 (Actual)
Dates: Start 2013-08-12 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2028-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Matt Ehrhardt, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (6):
- United States (6):
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - St. Jude Midwest Affiliate, Peoria, Illinois
  - Maine Children's Cancer Program (MCCP), Scarborough, Maine
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Harvard Cancer Center, Boston, Massachusetts
  - St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- [Derived] Castellino SM, Giulino-Roth L, Harker-Murray P, Kahn JM, Forlenza C, Cho S, Hoppe B, Parsons SK, Kelly KM; COG Hodgkin Lymphoma Committee. Children's Oncology Group's 2023 blueprint for research: Hodgkin lymphoma. Pediatr Blood Cancer. 2023 Sep;70 Suppl 6(Suppl 6):e30580. doi: 10.1002/pbc.30580. Epub 2023 Jul 28. PMID 37505794
- [Derived] Metzger ML, Link MP, Billett AL, Flerlage J, Lucas JT Jr, Mandrell BN, Ehrhardt MJ, Bhakta N, Yock TI, Friedmann AM, de Alarcon P, Luna-Fineman S, Larsen E, Kaste SC, Shulkin B, Lu Z, Li C, Hiniker SM, Donaldson SS, Hudson MM, Krasin MJ. Excellent Outcome for Pediatric Patients With High-Risk Hodgkin Lymphoma Treated With Brentuximab Vedotin and Risk-Adapted Residual Node Radiation. J Clin Oncol. 2021 Jul 10;39(20):2276-2283. doi: 10.1200/JCO.20.03286. Epub 2021 Apr 7. PMID 33826362
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 5 institutions between August 2013 to July 2018.
Pre-assignment Details: All the 77 patients are eligible for the study. Two out of 77 enrolled patients did not complete the study. One patient died during therapy, and 1 patient withdrew from the study. But both patients are evaluable for the primary objective.
Groups:
- AEPA/CAPDac: Ann Arbor stage IIB, IIIB, IVA, or IVB participants receive:
  2 cycles of AEPA chemotherapy:
  (A) Brentuximab vedotin 1.2 mg/kg IV (intravenous) days 1, 8 and 15, (E) Etoposide 125 mg/m^2 IV days 1-5, (P) Prednisone 60 mg/m^2/day PO (orally) days 1-15, (A) Doxorubicin 40 mg/m^2 IV days 1 and 15),
  Followed by 4 cycles of CAPDac:
  (C) Cyclophosphamide 500 mg/m^2 IV days 1 and 8, (A) Brentuximab vedotin 1.2 mg/kg IV days 1 and 8, (P) Prednisone 40 mg/m^2/day PO days 1-15, (Dac) Dacarbazine 250 mg/m^2 IV days 1-3.).
  Filgrastim 5 mcg/kg subcutaneous (SC) as clinically indicated.
  For those with lymph nodes that do not go into remission after 2 courses of AEPA chemotherapy, radiation therapy is given.
Period: Overall Study
Arm/Group | AEPA/CAPDac
Started | 77
Completed | 75
Not Completed | 2
Not completed — Death | 1
Not completed — Withdrawal of consent | 1

BASELINE CHARACTERISTICS:
Population: For staging: B symptoms (unexplained fevers, drenching night sweats or > 10% weight loss). A= absence of B symptoms
Arm/Group | AEPA/CAPDac
Number analyzed (Participants) | 77
Age, Continuous [Median (Full Range); unit: years] | 16 [6 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4
  Black or African American | 17
  White | 50
  More than one race | 4
  Others | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States: St. Jude Children's Research Hospital | 59
  United States: Stanford University Medical Center | 9
  United States: Dana Farber Cancer Institute | 4
  United States: Maine Medical Center | 1
  United States: Massachusetts General Hospital | 2
  United States: St. Jude Midwest Affiliate | 2
Histology [Count of Participants; unit: Participants] — Abbreviation: NOS, not otherwise specified.
  Participants
    Nodular sclerosing | 59
    Classical, NOS | 11
    Lymphocyte rich | 4
    Mixed cellularity | 3
Stage [Count of Participants; unit: Participants] — II: Involvement of 2 or more lymph node regions on the same side of the diaphragm (II) or localized contiguous involvement of a single extra-lymphatic organ or site and its regional lymph node(s) III: Involvement of lymph node regions on both sides of the diaphragm (III), which may also be accompanied by localized contiguous involvement of an extra-lymphatic organ or site (IIIE) IV: Disseminated (multifocal) involvement of 1 or more extra-lymphatic organs or tissues, with/without associated lymph node involvement, or isolated extra-lymphatic organ involvement with distant nodal involvement
  Participants
    IIB | 13
    IIIB | 19
    IVA | 12
    IVB | 33

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Initially Enrolled Patients That Have a Complete Response at Early Response Assessment Compared to Historical Control
Description: To determine the efficacy of 2 cycles of AEPA chemotherapy, the response rate for the first 32 evaluable participants enrolled was evaluated. If it shown efficacy (detect 20% increase complete rate with 80% power and 5% type I error compared with the proportion of historical control of HOD99 (NCT00145600) unfavorable risk patients had complete rate at week 8 of 17% (24/141), the response results will be reported in a national/international meeting and the study will continue to enroll for a total of 77 patients.
Time Frame: After the first 2 cycles of chemotherapy (at approximately 2 months after enrollment)
Population: The first 32 evaluable participants enrolled was evaluated.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- AEPA Chemotherapy: Ann Arbor stage IIB, IIIB, IVA, or IVB risk participants receive 2 cycles of AEPA chemotherapy (brentuximab vedotin, etoposide, prednisone, doxorubicin)
Arm/Group | AEPA Chemotherapy
Number analyzed (Participants) | 32
percentage of participants | 31.25 [18.04 to 47.21]
Statistical Analysis 1: Comparison: AEPA Chemotherapy; In the historical control (HOD99) 17% of patients had CR at week 8. Sample size for this objective is calculated based on a binomial distribution to test H0: p=17% vs. Ha: p>17%, where p is the true CR rate after 2 cycles of AEPA. 32 patients are needed to detect 20% increase of CR rate with 80% power and 5% type I error. If it shows efficacy, the response results will be reported, and the study will continue to enroll for a total of 77 patients to assess response and EFS; Test type: Superiority; The comparison of the complete rate between the first 32 evaluable participants and the historical control of HOD99 unfavorable risk patients was estimated by the binomial proportions test; Binomial proportions = 31.25

2. Primary Outcome: Percentage of Initially Enrolled Patients That Have a Complete Response at Early Response Assessment Compared to Historical Control
Description: To determine the efficacy of 2 cycles of AEPA chemotherapy, the response rate for the first 32 evaluable participants enrolled was evaluated. If it shown efficacy (detect 20% increase complete rate with 80% power and 5% type I error compared with the proportion of historical control of HOD99 unfavorable risk patients had complete rate at week 8 of 17% (24/141), the response results will be reported in a national/international meeting and the study will continue to enroll for a total of 77 patients.
Time Frame: After the first 2 cycles of chemotherapy (at approximately 2 months after enrollment)
Population: The first 32 evaluable participants enrolled was evaluated.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AEPA Chemotherapy
Number analyzed (Participants) | 32
percentage of participants | 31.25 [16.12 to 50.01]

3. Primary Outcome: Complete Response Rate Estimate for All Evaluable Participants
Description: To evaluate the safety of AEPA/CAPDac, as well as the efficacy (early complete response) after 2 cycles of AEPA chemotherapy in high-risk patients with Hodgkin Lymphoma (HL).
Time Frame: After the first 2 cycles of chemotherapy (at 2 months from enrollment for each participant)
Population: All the evaluable participants that completed the first 2 cycles of chemotherapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AEPA/CAPDac
Number analyzed (Participants) | 77
percentage of participants | 35 [24 to 46]
Statistical Analysis 1: Comparison: AEPA/CAPDac; Comparison of proportion of patient's complete response rate between HLHR13 and HOD99 (NCT00145600) unfavorable risk arm 2 (UR2); Test type: Superiority; p = 0.004, Fisher Exact

4. Primary Outcome: Comparison of the Event-free (EFS) Survival in High Risk HL Patients Treated With AEPA/CAPDac to the Historical Control HOD99 Unfavorable Risk 2 Arm (UR2).
Description: Event-free survival (EFS) is defined as the probability of survival between the date of study enrollment to the date of first event (relapsed or progressive disease, second malignancy, or death from any cause) or to last follow-up for patients without events. Under the proportional hazard model assumption, the two-sample log-rank test used to compare the EFS between HLHR13 and historical control of HOD99 unfavorable risk 2 arm (UR2).
Time Frame: From start of therapy to 2 years after completion of therapy (up to 3 years after study enrollment)
Population: For HLHR13, all the evaluable participants that treated with AEPA/CAPDac; for HOD99 Unfavorable Risk 2 Arm (UR2), all the evaluable participants that treated with Stanford V + RT.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | AEPA/CAPDac
Number analyzed (Participants) | 77
probability | 0.974 [0.951 to 0.997]
Statistical Analysis 1: Comparison: AEPA/CAPDac; The comparison of the EFS between HLHR13 and historical control of HOD99 unfavorable risk 2 arm (UR2) was done by the two-sample log-rank test; Test type: Superiority; p = 0.0008, Log Rank

5. Secondary Outcome: Local Failure Rate in High Risk HL Patients Treated With AEPA/CAPDac.
Description: The local failure rate within the high-risk HL participants treated with AEPA/CAPDac will be estimated with a 95% confidence interval using appropriate methods (e.g., estimate cumulative incidence in the presence of competing risks).
Time Frame: From start of therapy to 2 years after completion of therapy (up to 3 years after study enrollment)
Population: All the evaluable participants treated with AEPA/CAPDac.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | AEPA/CAPDac
Number analyzed (Participants) | 77
Probability | 0.013 [0.0003 to 0.0702]

6. Secondary Outcome: Descriptive of Hematological Adverse Events
Description: To describe acute hematologic, neuropathic, and infectious toxicities as they relate to transfusion requirements, growth factor support, episodes of febrile neutropenia and hospitalizations, according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 4.0.
Time Frame: From enrollment to end of therapy (approximately 8 months)
Population: Toxicities reported below for the current study (HLHR13) include all reported hematological toxicities from a participant's on-study date through end of therapy.
Measure: Count of Participants; unit: Participants
Groups:
- Cycle 1 - Grade 2; Cycle 1 - Grade 3-4; Cycle 2 - Grade 2; Cycle 2 - Grade 3-4: Participants receive AEPA regimen for 2 cycles (cycle length 28 days)
  (A) Brentuximab vedotin 1.2 mg/kg IV (E) Etoposide 125 mg/m^2 IV (P) Prednisone 60 mg/m^2/day PO (orally) (A) Doxorubicin 40 mg/m^2 IV
  For those with lymph nodes that do not go into remission after 2 courses of AEPA chemotherapy, radiation therapy will be given.
- Cycle 3 - Grade 2; Cycle 3 - Grade 3-4; Cycle 4 - Grade 2; Cycle 4 - Grade 3-4; Cycle 5 - Grade 2; Cycle 5 - Grade 3-4; Cycle 6 - Grade 2; Cycle 6 - Grade 3-4: Participants receive CAPDac regimen for 4 cycles (cycle length 21 days):
  (C) Cyclophosphamide IV 500 mg/m^2 (A) Brentuximab vedotin 1.2 mg/kg IV (P) Prednisone 40 mg/40 mg/m^2/day PO (Dac) Dacarbazine 250 mg/m^2 IV
Arm/Group | Cycle 1 - Grade 2 | Cycle 1 - Grade 3-4 | Cycle 2 - Grade 2 | Cycle 2 - Grade 3-4 | Cycle 3 - Grade 2 | Cycle 3 - Grade 3-4 | Cycle 4 - Grade 2 | Cycle 4 - Grade 3-4 | Cycle 5 - Grade 2 | Cycle 5 - Grade 3-4 | Cycle 6 - Grade 2 | Cycle 6 - Grade 3-4
Number analyzed (Participants) | 77 | 77 | 77 | 77 | 77 | 77 | 76 | 76 | 76 | 76 | 76 | 76
Participants
  Leukopenia | 15 | 49 | 28 | 23 | 8 | 4 | 5 | 5 | 7 | 2 | 14 | 5
  Neutropenia | 5 | 62 | 13 | 51 | 7 | 10 | 5 | 3 | 4 | 3 | 8 | 6
  Lymphopenia | 15 | 36 | 18 | 15 | 9 | 7 | 16 | 15 | 13 | 22 | 20 | 31
  Anemia | 23 | 12 | 28 | 5 | 6 | 1 | 6 | 0 | 4 | 1 | 2 | 1
  Thrombocytopenia | 3 | 3 | 2 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 2

7. Secondary Outcome: Descriptive of Infectious Adverse Events
Description: as for outcome 6
Time Frame: From enrollment to end of therapy (approximately 8 months)
Population: Toxicities reported below for the current study (HLHR13) include all reported infectious toxicities from a participant's on-study date through end of therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Cycle 1 - Grade 2 | Cycle 1 - Grade 3-4 | Cycle 2 - Grade 2 | Cycle 2 - Grade 3-4 | Cycle 3 - Grade 2 | Cycle 3 - Grade 3-4 | Cycle 4 - Grade 2 | Cycle 4 - Grade 3-4 | Cycle 5 - Grade 2 | Cycle 5 - Grade 3-4 | Cycle 6 - Grade 2 | Cycle 6 - Grade 3-4
Number analyzed (Participants) | 77 | 77 | 77 | 77 | 77 | 77 | 76 | 76 | 76 | 76 | 76 | 76
Participants
  Febrile neutropenia | 0 | 6 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
  Mucositis | 10 | 2 | 6 | 4 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
  Upper respiratory infection | 5 | 2 | 3 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Genitourinary infection | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0

8. Secondary Outcome: Descriptive of Neuropathic Adverse Events
Description: as for outcome 6
Time Frame: From enrollment to end of therapy (approximately 8 months)
Population: Toxicities reported below for the current study (HLHR13) include all reported neuropathic toxicities from a participant's on-study date through end of therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Cycle 1 - Grade 2 | Cycle 1 - Grade 3-4 | Cycle 2 - Grade 2 | Cycle 2 - Grade 3-4 | Cycle 3 - Grade 2 | Cycle 3 - Grade 3-4 | Cycle 4 - Grade 2 | Cycle 4 - Grade 3-4 | Cycle 5 - Grade 2 | Cycle 5 - Grade 3-4 | Cycle 6 - Grade 2 | Cycle 6 - Grade 3-4
Number analyzed (Participants) | 77 | 77 | 77 | 77 | 77 | 77 | 76 | 76 | 76 | 76 | 76 | 76
Participants
  Peripheral sensory neuropathy | 0 | 0 | 1 | 0 | 2 | 0 | 3 | 0 | 1 | 0 | 1 | 0
  Pain in extremity | 3 | 1 | 4 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0
  Neuralgia | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Pain NOS | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

9. Secondary Outcome: To Assess the Patient Reported Symptoms and Health-related Quality of Life in Children With High Risk HL Compared to Those Treated on the Unfavorable HOD99 Treatment Arm (UR2) at Multiple Time Points. (PedsQL v.3.0)
Description: Assess and compare the patient reported quality of life and symptom distress to that of patients treated on the HOD99 unfavorable risk 2 arm (UR2) using the Peds Quality of Life version 3. The QL scoring is a 5-point Likert scale from 0 (never) to 4 (almost always). Scores are transformed on a scale from 0 to 100. Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. Total score is the sum of all items over the number of items answered on all scales. For both the total score and subscales the range is 0-100. The total score is the sum of all items from each subscale, over the number of items answered on the scale. The total score is the sum of all items on the scale over the number of items answer. If >50% of the items are missing the score should not be computed. If >50% are completed, impute the mean of the completed items in a scale. The Higher the score the better quality of life.
Time Frame: At Diagnosis (baseline) (T1), completion of 2 cycles of chemotherapy (approximately 2 months) (T2), completion of 4 cycles of chemotherapy (approximately 4 months) (T3), completion of radiation (approximately 8 months) (T4)
Population: Each institution made the decision whether to complete the QoL objective. Participation in the Quality of Life part of the trial is voluntary for participating institutions and voluntary by patient. The Peds QL 3.0 data was not collected on the HOD 99 patients at the T1 time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- AEPA/CAPDac: Ann Arbor stage IIB, IIIB, IVA, or IVB risk participants received 2 cycles of AEPA/CAPDac chemotherapy and reported symptoms distress scale (SDS).
- HOD99 Unfavorable Risk 2 Arm (UR2): Ann Arbor stage IIB, IIIB, or any IV risk participants received 12 weeks Stanford V Chemotherapy
Arm/Group | AEPA/CAPDac | HOD99 Unfavorable Risk 2 Arm (UR2)
Number analyzed (Participants) | 77 | 146
score on a scale
  PedsQL v.3.0 Total Score-T1: number analyzed (Participants) | 63 | 0
  PedsQL v.3.0 Total Score-T1 | 73.38 (15.97) |
  PedsQL v.3.0 Total Score-T2: number analyzed (Participants) | 62 | 85
  PedsQL v.3.0 Total Score-T2 | 80.41 (14.68) | 71.92 (14.58)
  PedsQL v.3.0 Total Score-T3: number analyzed (Participants) | 58 | 76
  PedsQL v.3.0 Total Score-T3 | 83.33 (13.87) | 73.78 (17.72)
  PedsQL v.3.0 Total Score-T4: number analyzed (Participants) | 50 | 62
  PedsQL v.3.0 Total Score-T4 | 85.33 (13.62) | 79.92 (16.25)
  PedsQL v.3.0 Pain and Hurt-T1: number analyzed (Participants) | 63 | 0
  PedsQL v.3.0 Pain and Hurt-T1 | 73.41 (27.45) |
  PedsQL v.3.0 Pain and Hurt-T2: number analyzed (Participants) | 62 | 87
  PedsQL v.3.0 Pain and Hurt-T2 | 71.77 (29.94) | 66.09 (27.49)
  PedsQL v.3.0 Pain and Hurt-T3: number analyzed (Participants) | 58 | 77
  PedsQL v.3.0 Pain and Hurt-T3 | 72.63 (30.03) | 69.81 (29.34)
  PedsQL v.3.0 Pain and Hurt-T4: number analyzed (Participants) | 50 | 66
  PedsQL v.3.0 Pain and Hurt-T4 | 77.5 (30.3) | 82.2 (25.39)
  PedsQL v.3.0 Nausea-T1: number analyzed (Participants) | 63 | 0
  PedsQL v.3.0 Nausea-T1 | 73.97 (21.2) |
  PedsQL v.3.0 Nausea-T2: number analyzed (Participants) | 62 | 87
  PedsQL v.3.0 Nausea-T2 | 75.52 (23.92) | 60.5 (23.83)
  PedsQL v.3.0 Nausea-T3: number analyzed (Participants) | 58 | 77
  PedsQL v.3.0 Nausea-T3 | 79.66 (20.73) | 60.26 (26.92)
  PedsQL v.3.0 Nausea-T4: number analyzed (Participants) | 50 | 64
  PedsQL v.3.0 Nausea-T4 | 88.1 (17.67) | 78.13 (22.69)
  PedsQL v.3.0 Procedural Anxiety-T1: number analyzed (Participants) | 63 | 0
  PedsQL v.3.0 Procedural Anxiety-T1 | 58.6 (37) |
  PedsQL v.3.0 Procedural Anxiety-T2: number analyzed (Participants) | 62 | 87
  PedsQL v.3.0 Procedural Anxiety-T2 | 77.55 (26.64) | 71.17 (27.72)
  PedsQL v.3.0 Procedural Anxiety-T3: number analyzed (Participants) | 58 | 76
  PedsQL v.3.0 Procedural Anxiety-T3 | 81.61 (24.47) | 73.46 (27.98)
  PedsQL v.3.0 Procedural Anxiety-T4: number analyzed (Participants) | 50 | 66
  PedsQL v.3.0 Procedural Anxiety-T4 | 76.83 (30.36) | 77.65 (24.2)
  PedsQL v.3.0 Treatment Anxiety-T1: number analyzed (Participants) | 63 | 0
  PedsQL v.3.0 Treatment Anxiety-T1 | 84.52 (21.47) |
  PedsQL v.3.0 Treatment Anxiety-T2: number analyzed (Participants) | 61 | 87
  PedsQL v.3.0 Treatment Anxiety-T2 | 91.39 (14.67) | 85.92 (17.06)
  PedsQL v.3.0 Treatment Anxiety-T3: number analyzed (Participants) | 58 | 77
  PedsQL v.3.0 Treatment Anxiety-T3 | 93.97 (12.37) | 85.06 (23.11)
  PedsQL v.3.0 Treatment Anxiety-T4: number analyzed (Participants) | 50 | 66
  PedsQL v.3.0 Treatment Anxiety-T4 | 93.17 (13.95) | 83.71 (22.9)
  PedsQL v.3.0 Worry-T1: number analyzed (Participants) | 62 | 0
  PedsQL v.3.0 Worry-T1 | 69.22 (24.08) |
  PedsQL v.3.0 Worry-T2: number analyzed (Participants) | 62 | 86
  PedsQL v.3.0 Worry-T2 | 77.55 (22.51) | 64.63 (25.01)
  PedsQL v.3.0 Worry-T3: number analyzed (Participants) | 58 | 77
  PedsQL v.3.0 Worry-T3 | 84.2 (17.01) | 66.45 (25.33)
  PedsQL v.3.0 Worry-T4: number analyzed (Participants) | 50 | 66
  PedsQL v.3.0 Worry-T4 | 82.17 (20.89) | 69.57 (29.58)
  PedsQL v.3.0 Cognitive Problems-T1: number analyzed (Participants) | 63 | 0
  PedsQL v.3.0 Cognitive Problems-T1 | 72.34 (23.09) |
  PedsQL v.3.0 Cognitive Problems-T2: number analyzed (Participants) | 62 | 86
  PedsQL v.3.0 Cognitive Problems-T2 | 81.25 (21.06) | 75.72 (19.48)
  PedsQL v.3.0 Cognitive Problems-T3: number analyzed (Participants) | 58 | 77
  PedsQL v.3.0 Cognitive Problems-T3 | 84.38 (19.41) | 78.38 (22.03)
  PedsQL v.3.0 Cognitive Problems-T4: number analyzed (Participants) | 49 | 65
  PedsQL v.3.0 Cognitive Problems-T4 | 87.04 (18.95) | 81.69 (17.84)
  PedsQL v.3.0 Perceived Physical Appearance-T1: number analyzed (Participants) | 61 | 0
  PedsQL v.3.0 Perceived Physical Appearance-T1 | 79.64 (25.21) |
  PedsQL v.3.0 Perceived Physical Appearance-T2: number analyzed (Participants) | 62 | 87
  PedsQL v.3.0 Perceived Physical Appearance-T2 | 83.53 (22.99) | 78.07 (24.91)
  PedsQL v.3.0 Perceived Physical Appearance-T3: number analyzed (Participants) | 58 | 77
  PedsQL v.3.0 Perceived Physical Appearance-T3 | 82.69 (22.29) | 79.87 (22.47)
  PedsQL v.3.0 Perceived Physical Appearance-T4: number analyzed (Participants) | 50 | 64
  PedsQL v.3.0 Perceived Physical Appearance-T4 | 85.17 (22.48) | 79.95 (23.79)
  PedsQL v.3.0 Communication-T1: number analyzed (Participants) | 62 | 0
  PedsQL v.3.0 Communication-T1 | 74.6 (27.3) |
  PedsQL v.3.0 Communication-T2: number analyzed (Participants) | 61 | 87
  PedsQL v.3.0 Communication-T2 | 85.38 (20.73) | 79.02 (18.58)
  PedsQL v.3.0 Communication-T3: number analyzed (Participants) | 58 | 77
  PedsQL v.3.0 Communication-T3 | 85.34 (20.9) | 81.93 (21.22)
  PedsQL v.3.0 Communication-T4: number analyzed (Participants) | 50 | 64
  PedsQL v.3.0 Communication-T4 | 87.33 (17.6) | 84.24 (21.16)
Statistical Analysis 1: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Total Score-T2, completion of 2 cycles of chemotherapy (approximately 2 months); Test type: Superiority; p < .001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Total Score-T3, completion of 4 cycles of chemotherapy (approximately 4 months); Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Total Score-T4, completion of radiation (approximately 8 months); Test type: Superiority; p = 0.067, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Pain and Hurt-T2, completion of 2 cycles of chemotherapy (approximately 2 months); Test type: Superiority; p = 0.115, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Pain and Hurt-T3, completion of 4 cycles of chemotherapy (approximately 4 months); Test type: Superiority; p = 0.455, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Pain and Hurt-T4, completion of radiation (approximately 8 months); Test type: Superiority; p = 0.636, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Nausea-T2, completion of 2 cycles of chemotherapy (approximately 2 months); Test type: Superiority; p < .001, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Nausea-T3, completion of 4 cycles of chemotherapy (approximately 4 months); Test type: Superiority; p < .001, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Nausea-T4, completion of radiation (approximately 8 months); Test type: Superiority; p = 0.006, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Procedural Anxiety-T2, completion of 2 cycles of chemotherapy (approximately 2 months); Test type: Superiority; p = 0.099, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Procedural Anxiety-T3, completion of 4 cycles of chemotherapy (approximately 4 months); Test type: Superiority; p = 0.050, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Procedural Anxiety-T4, completion of radiation (approximately 8 months); Test type: Superiority; p = 0.520, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Treatment Anxiety-T2, completion of 2 cycles of chemotherapy (approximately 2 months); Test type: Superiority; p = 0.024, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Treatment Anxiety-T3, completion of 4 cycles of chemotherapy (approximately 4 months); Test type: Superiority; p = 0.011, Wilcoxon (Mann-Whitney)
Statistical Analysis 15: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Treatment Anxiety-T4, completion of radiation (approximately 8 months); Test type: Superiority; p = 0.009, Wilcoxon (Mann-Whitney)
Statistical Analysis 16: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Worry-T2, completion of 2 cycles of chemotherapy (approximately 2 months); Test type: Superiority; p < .001, Wilcoxon (Mann-Whitney)
Statistical Analysis 17: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Worry-T3, completion of 4 cycles of chemotherapy (approximately 4 months); Test type: Superiority; p < .001, Wilcoxon (Mann-Whitney)
Statistical Analysis 18: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Worry-T4, completion of radiation (approximately 8 months); Test type: Superiority; p = 0.035, Wilcoxon (Mann-Whitney)
Statistical Analysis 19: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Cognitive Problems-T2, completion of 2 cycles of chemotherapy (approximately 2 months); Test type: Superiority; p = 0.037, Wilcoxon (Mann-Whitney)
Statistical Analysis 20: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Cognitive Problems-T3, completion of 4 cycles of chemotherapy (approximately 4 months); Test type: Superiority; p = 0.043, Wilcoxon (Mann-Whitney)
Statistical Analysis 21: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Cognitive Problems-T4, completion of radiation (approximately 8 months); Test type: Superiority; p = 0.044, Wilcoxon (Mann-Whitney)
Statistical Analysis 22: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Perceived Physical Appearance-T2, completion of 2 cycles of chemotherapy (approximately 2 months); Test type: Superiority; p = 0.091, Wilcoxon (Mann-Whitney)
Statistical Analysis 23: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Perceived Physical Appearance-T3, completion of 4 cycles of chemotherapy (approximately 4 months); Test type: Superiority; p = 0.248, Wilcoxon (Mann-Whitney)
Statistical Analysis 24: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Perceived Physical Appearance-T4, completion of radiation (approximately 8 months); Test type: Superiority; p = 0.069, Wilcoxon (Mann-Whitney)
Statistical Analysis 25: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Communication-T2, completion of 2 cycles of chemotherapy (approximately 2 months); Test type: Superiority; p = 0.010, Wilcoxon (Mann-Whitney)
Statistical Analysis 26: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Communication-T3, completion of 4 cycles of chemotherapy (approximately 4 months); Test type: Superiority; p = 0.292, Wilcoxon (Mann-Whitney)
Statistical Analysis 27: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.3.0 Communication-T4, completion of radiation (approximately 8 months); Test type: Superiority; p = 0.429, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: To Assess the Patient Reported Symptoms and Health-related Quality of Life in Children With High Risk HL Compared to Those Treated on the Unfavorable HOD99 Treatment Arm (UR2) at Multiple Time Points. (PedsQL v.4.0)
Description: Assess and compare the patient reported quality of life and symptom distress to that of patients treated on the HOD99 unfavorable risk 2 arm (UR2) using the Peds Quality of Life version 4. The QL scoring is a 5-point Likert scale from 0 (never) to 4 (almost always). Scores are transformed on a scale from 0 to 100. Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. Total score is the sum of all items over the number of items answered on all scales. For both the total score and subscales the range is 0-100. The total score is the sum of all items from each subscale, over the number of items answered on the scale. The total score is the sum of all items on the scale over the number of items answer. If >50% of the items are missing the score should not be computed. If >50% are completed, impute the mean of the completed items in a scale. The Higher the score the better quality of life.
Time Frame: as for outcome 9
Population: Each institution made the decision whether to complete the QoL objective. Participation in the Quality of Life part of the trial is voluntary for participating institutions and voluntary by patient.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- AEPA/CAPDac: Ann Arbor stage IIB, IIIB, IVA, or IVB risk participants received 2 cycles of AEPE/CAPDac chemotherapy and reported symptoms distress scale (SDS).
Arm/Group | AEPA/CAPDac | HOD99 Unfavorable Risk 2 Arm (UR2)
Number analyzed (Participants) | 77 | 146
score on a scale
  PedsQL v.4.0 Total Score-T1: number analyzed (Participants) | 63 | 78
  PedsQL v.4.0 Total Score-T1 | 72.94 (17.63) | 72.48 (17.37)
  PedsQL v.4.0 Total Score-T2: number analyzed (Participants) | 62 | 76
  PedsQL v.4.0 Total Score-T2 | 79.38 (17.43) | 73.54 (16.71)
  PedsQL v.4.0 Total Score-T3: number analyzed (Participants) | 58 | 70
  PedsQL v.4.0 Total Score-T3 | 80.39 (14.96) | 77.68 (17.25)
  PedsQL v.4.0 Total Score-T4: number analyzed (Participants) | 52 | 59
  PedsQL v.4.0 Total Score-T4 | 86.06 (14.53) | 84.58 (15.02)
  PedsQL v.4.0 Physical Functioning-T1: number analyzed (Participants) | 63 | 85
  PedsQL v.4.0 Physical Functioning-T1 | 69.54 (21.78) | 70.41 (26.09)
  PedsQL v.4.0 Physical Functioning-T2: number analyzed (Participants) | 62 | 88
  PedsQL v.4.0 Physical Functioning-T2 | 73.86 (24.14) | 70.06 (22.73)
  PedsQL v.4.0 Physical Functioning-T3: number analyzed (Participants) | 58 | 79
  PedsQL v.4.0 Physical Functioning-T3 | 74.02 (22.13) | 72.94 (25.25)
  PedsQL v.4.0 Physical Functioning-T4: number analyzed (Participants) | 52 | 66
  PedsQL v.4.0 Physical Functioning-T4 | 82.45 (23.24) | 83.57 (18.86)
  PedsQL v.4.0 Emotional Functioning-T1: number analyzed (Participants) | 63 | 85
  PedsQL v.4.0 Emotional Functioning-T1 | 71.75 (24.38) | 67.18 (18.25)
  PedsQL v.4.0 Emotional Functioning-T2: number analyzed (Participants) | 62 | 88
  PedsQL v.4.0 Emotional Functioning-T2 | 83.06 (16.63) | 71.31 (20.96)
  PedsQL v.4.0 Emotional Functioning-T3: number analyzed (Participants) | 58 | 79
  PedsQL v.4.0 Emotional Functioning-T3 | 82.07 (18.43) | 75.06 (22.38)
  PedsQL v.4.0 Emotional Functioning-T4: number analyzed (Participants) | 52 | 66
  PedsQL v.4.0 Emotional Functioning-T4 | 84.81 (19.75) | 80.87 (20.63)
  PedsQL v.4.0 Social Functioning-T1: number analyzed (Participants) | 63 | 85
  PedsQL v.4.0 Social Functioning-T1 | 86.21 (17.05) | 86.22 (17.69)
  PedsQL v.4.0 Social Functioning-T2: number analyzed (Participants) | 62 | 88
  PedsQL v.4.0 Social Functioning-T2 | 88.47 (15.85) | 86.82 (15.42)
  PedsQL v.4.0 Social Functioning-T3: number analyzed (Participants) | 58 | 79
  PedsQL v.4.0 Social Functioning-T3 | 90.22 (12.41) | 88.86 (13.84)
  PedsQL v.4.0 Social Functioning-T4: number analyzed (Participants) | 52 | 66
  PedsQL v.4.0 Social Functioning-T4 | 92.31 (11.57) | 91.44 (14.35)
  PedsQL v.4.0 School Functioning-T1: number analyzed (Participants) | 61 | 78
  PedsQL v.4.0 School Functioning-T1 | 65.49 (22.72) | 67.82 (19.65)
  PedsQL v.4.0 School Functioning-T2: number analyzed (Participants) | 61 | 76
  PedsQL v.4.0 School Functioning-T2 | 75.66 (24.66) | 66.91 (21.79)
  PedsQL v.4.0 School Functioning-T3: number analyzed (Participants) | 56 | 70
  PedsQL v.4.0 School Functioning-T3 | 79.2 (21.49) | 69.1 (24.27)
  PedsQL v.4.0 School Functioning-T4: number analyzed (Participants) | 50 | 59
  PedsQL v.4.0 School Functioning-T4 | 86.9 (18.62) | 79.32 (17.77)
Statistical Analysis 1: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.4.0 Total Score-T1, At Diagnosis (baseline); Test type: Superiority; p = 0.975, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.4.0 Total Score-T2, completion of 2 cycles of chemotherapy (approximately 2 months); Test type: Superiority; p = 0.032, t-test, 2 sided
Statistical Analysis 3: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.4.0 Total Score-T3, completion of 4 cycles of chemotherapy (approximately 4 months); Test type: Superiority; p = 0.497, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.4.0 Total Score-T4, completion of radiation (approximately 8 months); Test type: Superiority; p = 0.399, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.4.0 Physical Functioning-T1, At Diagnosis (baseline); Test type: Superiority; p = 0.451, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.4.0 Physical Functioning-T2, completion of 2 cycles of chemotherapy (approximately 2 months); Test type: Superiority; p = 0.198, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.4.0 Physical Functioning-T3, completion of 4 cycles of chemotherapy (approximately 4 months); Test type: Superiority; p = 0.967, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.4.0 Physical Functioning-T4, completion of radiation (approximately 8 months); Test type: Superiority; p = 0.647, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.4.0 Emotional Functioning-T1, At Diagnosis (baseline); Test type: Superiority; p = 0.145, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.4.0 Emotional Functioning-T2, completion of 2 cycles of chemotherapy (approximately 2 months); Test type: Superiority; p < .001, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.4.0 Emotional Functioning-T3, completion of 4 cycles of chemotherapy (approximately 4 months); Test type: Superiority; p = 0.073, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.4.0 Emotional Functioning-T4, completion of radiation (approximately 8 months); Test type: Superiority; p = 0.156, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.4.0 Social Functioning-T1, At Diagnosis (baseline); Test type: Superiority; p = 0.844, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.4.0 Social Functioning-T2, completion of 2 cycles of chemotherapy (approximately 2 months); Test type: Superiority; p = 0.206, Wilcoxon (Mann-Whitney)
Statistical Analysis 15: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.4.0 Social Functioning-T3, completion of 4 cycles of chemotherapy (approximately 4 months); Test type: Superiority; p = 0.491, Wilcoxon (Mann-Whitney)
Statistical Analysis 16: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.4.0 Social Functioning-T4, completion of radiation (approximately 8 months); Test type: Superiority; p = 0.906, Wilcoxon (Mann-Whitney)
Statistical Analysis 17: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.4.0 School Functioning-T1, At Diagnosis (baseline); Test type: Superiority; p = 0.580, Wilcoxon (Mann-Whitney)
Statistical Analysis 18: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.4.0 School Functioning-T2, completion of 2 cycles of chemotherapy (approximately 2 months); Test type: Superiority; p = 0.012, Wilcoxon (Mann-Whitney)
Statistical Analysis 19: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.4.0 School Functioning-T3, completion of 4 cycles of chemotherapy (approximately 4 months); Test type: Superiority; p = 0.010, Wilcoxon (Mann-Whitney)
Statistical Analysis 20: Comparison: AEPA/CAPDac vs HOD99 Unfavorable Risk 2 Arm (UR2); PedsQL v.4.0 School Functioning-T4, completion of radiation (approximately 8 months); Test type: Superiority; p = 0.005, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Response Rate
Description: Response compared to the Euro-Net C1 after 2 cycles of AEPA.
Time Frame: after the first 2 cycles of chemotherapy (at approximately 2 months after enrollment)
Reporting Status: Not Posted

12. Secondary Outcome: Patient Quality of Life (QoL)
Description: Patient QOL will be measured at multiple time points to assess the patient's physical emotional, social, and school functioning.
  The QL scoring is a 5-point Likert scale from 0 (never) to 4 (almost always). Scores are transformed on a scale from 0 to 100. Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. Total score is the sum of all items over the number of items answered on all scales. For both the total score and subscales the range is 0-100. The total score is the sum of all items from each subscale, over the number of items answered on the scale. The total score is the sum of all items on the scale over the number of items answer. If >50% of the items are missing the score should not be computed. If >50% are completed, impute the mean of the completed items in a scale. The Higher the score the better quality of life.
Time Frame: At various time points from diagnosis through 5 years off therapy. (up to approximately 6 years from enrollment).
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Timepoint 1 (T1): At Diagnosis (baseline)
- Timepoint 4 (T4): Course 2 Day 1
- Timepoint 6 (T6): Course 3 Day 1
- Timepoint 8 (T8): Course 6 Day 1
- Timepoint 10 (T10): 4-6 weeks after chemotherapy or 4-6 weeks after radiation
- Timepoint 11 (T11): 1 year off therapy
- Timepoint 12 (T12): 2 years off therapy (approximately 2 years and 8 months
- Timepoint 13 (T13): 5 years off therapy (approximately 5 years and 8 months)
Arm/Group | Timepoint 1 (T1) | Timepoint 4 (T4) | Timepoint 6 (T6) | Timepoint 8 (T8) | Timepoint 10 (T10) | Timepoint 11 (T11) | Timepoint 12 (T12) | Timepoint 13 (T13)
Number analyzed (Participants) | 63 | 64 | 62 | 58 | 52 | 51 | 39 | 35
score on a scale
  Physical Functioning | 69.5 (21.8) | 75.8 (21.8) | 73.9 (24.1) | 74 (22.1) | 82.5 (23.2) | 87.7 (20.3) | 87.1 (20.7) | 88.8 (19.4)
  Emotional Functioning | 71.7 (24.4) | 80.3 (20.2) | 83.1 (16.6) | 82.1 (18.4) | 84.8 (19.8) | 88.4 (18.8) | 88.2 (16.4) | 80.9 (22.8)
  Social Functioning: number analyzed (Participants) | 63 | 64 | 62 | 58 | 52 | 50 | 39 | 35
  Social Functioning | 86.2 (17) | 87.2 (18.3) | 88.5 (15.9) | 90.2 (12.4) | 92.3 (11.6) | 93.8 (11.9) | 94 (12.8) | 95.3 (12.2)
  School Functioning: number analyzed (Participants) | 61 | 58 | 61 | 56 | 50 | 50 | 39 | 35
  School Functioning | 65.5 (22.7) | 75.7 (24.3) | 75.7 (24.7) | 79.2 (21.5) | 86.9 (18.6) | 85.4 (16.2) | 87.2 (13.1) | 81.5 (23.1)

13. Secondary Outcome: Parent Proxy Quality of Life (QoL)
Description: Parent's assessment of child's physical, emotional, social and school functioning over multiple time points.
  The QL scoring is a 5-point Likert scale from 0 (never) to 4 (almost always). Scores are transformed on a scale from 0 to 100. Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. Total score is the sum of all items over the number of items answered on all scales. For both the total score and subscales the range is 0-100. The total score is the sum of all items from each subscale, over the number of items answered on the scale. The total score is the sum of all items on the scale over the number of items answer. If >50% of the items are missing the score should not be computed. If >50% are completed, impute the mean of the completed items in a scale. The Higher the score the better quality of life.
Time Frame: At various time points from diagnosis through 5 years off therapy. (up to approximately 6 years from enrollment)
Population: Each institution made the decision whether to complete the QoL objective. Participation in the Quality of Life part of the trial is voluntary for participating institutions and voluntary by parent.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Timepoint 1 (T1) | Timepoint 4 (T4) | Timepoint 6 (T6) | Timepoint 8 (T8) | Timepoint 10 (T10) | Timepoint 11 (T11) | Timepoint 12 (T12) | Timepoint 13 (T13)
Number analyzed (Participants) | 62 | 60 | 57 | 55 | 46 | 41 | 30 | 10
score on a scale
  Physical Functioning | 61.8 (26.9) | 65.3 (20.8) | 66.8 (22.3) | 65.6 (24.1) | 74.5 (25.6) | 76.6 (29.0) | 75 (26.4) | 84.7 (29.1)
  Emotional Functioning: number analyzed (Participants) | 62 | 59 | 57 | 55 | 46 | 41 | 30 | 10
  Emotional Functioning | 61.9 (23.1) | 69.3 (25.2) | 72 (22.5) | 73.7 (21.4) | 78.6 (21) | 84.2 (20.3) | 79 (23.3) | 85.5 (19.2)
  Social Functioning: number analyzed (Participants) | 62 | 59 | 56 | 55 | 46 | 41 | 30 | 10
  Social Functioning | 80.3 (18.8) | 79.2 (21.6) | 79.6 (18.4) | 79.2 (19.8) | 84.5 (20.1) | 87.8 (17.9) | 82.5 (22.8) | 92.6 (13.5)
  School Functioning: number analyzed (Participants) | 61 | 56 | 52 | 53 | 41 | 41 | 29 | 10
  School Functioning | 63.2 (25.4) | 68.5 (25.6) | 67.1 (25.3) | 70.5 (25.2) | 80.3 (21.7) | 82.2 (22.9) | 78.2 (22.5) | 81 (19.4)

14. Secondary Outcome: Correlation of Agreement Between Patient QoL and Parent Proxy QoL at Multiple Time Points
Description: The correlation of agreement between patient and parent Quality of Life is calculated by using the Pearson's Correlation Coefficient, which considers only the record with both parent and patient data.
  The QL scoring is a 5-point Likert scale from 0 (never) to 4 (almost always). Scores are transformed on a scale from 0 to 100. Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. Total score is the sum of all items over the number of items answered on all scales. For both the total score and subscales the range is 0-100. The total score is the sum of all items from each subscale, over the number of items answered on the scale. The total score is the sum of all items on the scale over the number of items answer. If >50% of the items are missing the score should not be computed. If >50% are completed, impute the mean of the completed items in a scale. The Higher the score the better quality of life.
Time Frame: At various time points from diagnosis through 5 years off therapy. (up to approximately 6 years from enrollment)
Population: Each institution made the decision whether to complete the QoL objective. Participation in the Quality of Life part of the trial is voluntary for participating institutions and voluntary by participant.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Timepoint 1 (T1) | Timepoint 4 (T4) | Timepoint 6 (T6) | Timepoint 8 (T8) | Timepoint 10 (T10) | Timepoint 11 (T11) | Timepoint 12 (T12) | Timepoint 13 (T13)
Number analyzed (Participants) | 62 | 60 | 56 | 54 | 45 | 41 | 30 | 10
correlation coefficient
  Physical Functioning | 0.701 [0.547 to 0.809] | 0.503 [0.286 to 0.671] | 0.536 [0.318 to 0.7] | 0.575 [0.363 to 0.73] | 0.406 [0.128 to 0.625] | 0.528 [0.263 to 0.719] | 0.468 [0.129 to 0.709] | 0.294 [-0.411 to 0.78]
  Social Functioning: number analyzed (Participants) | 62 | 59 | 56 | 54 | 45 | 41 | 30 | 10
  Social Functioning | 0.309 [0.064 to 0.518] | 0.566 [0.362 to 0.718] | 0.534 [0.313 to 0.7] | 0.242 [-0.028 to 0.479] | 0.086 [-0.213 to 0.371] | 0.327 [0.021 to 0.577] | 0.135 [-0.236 to 0.473] | -0.027 [-0.645 to 0.613]
  Emotional Functioning: number analyzed (Participants) | 62 | 59 | 55 | 54 | 45 | 41 | 30 | 10
  Emotional Functioning | 0.593 [0.402 to 0.734] | 0.664 [0.491 to 0.786] | 0.648 [0.464 to 0.778] | 0.588 [0.38 to 0.739] | 0.344 [0.056 to 0.579] | 0.671 [0.457 to 0.811] | 0.291 [-0.077 to 0.59] | 0.756 [0.24 to 0.939]
  School Functioning: number analyzed (Participants) | 62 | 53 | 51 | 51 | 40 | 41 | 29 | 10
  School Functioning | 0.444 [0.211 to 0.628] | 0.577 [0.364 to 0.733] | 0.501 [0.261 to 0.682] | 0.441 [0.188 to 0.639] | 0.694 [0.488 to 0.827] | 0.315 [0.004 to 0.57] | 0.209 [-0.17 to 0.535] | 0.574 [-0.088 to 0.884]

ADVERSE EVENTS:
Time Frame: Acute adverse events were collected from each participant's on-study date through the end of therapy, through study completion, an average of 1 year. The timeframe for All-Cause Mortality was from start of therapy to 2 years after completion of therapy (up to 3 years after study enrollment).
Arm/Group | AEPA/CAPDac
All-Cause Mortality (participants affected / at risk) | 1/77
Serious Adverse Events (participants affected / at risk) | 2/77
Other Adverse Events (participants affected / at risk) | 75/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AEPA/CAPDac (N=77)
Ventricular tachycardia (Cardiac disorders) | 1
Neutrophil count decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AEPA/CAPDac (N=77)
Neutrophil count decreased (Investigations) | 75
Lymphocyte count decreased (Investigations) | 74
White blood cell decreased (Investigations) | 73
Anemia (Blood and lymphatic system disorders) | 71
Alanine aminotransferase increased (Investigations) | 56
Weight gain (Investigations) | 55
Platelet count decreased (Investigations) | 51
Nausea (Gastrointestinal disorders) | 50
Hyperglycemia (Metabolism and nutrition disorders) | 39
Hypoalbuminemia (Metabolism and nutrition disorders) | 36
Vomiting (Gastrointestinal disorders) | 34
Aspartate aminotransferase increased (Investigations) | 28
Constipation (Gastrointestinal disorders) | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 25
Headache (Nervous system disorders) | 24
Mucositis oral (Gastrointestinal disorders) | 23
Hyponatremia (Metabolism and nutrition disorders) | 23
Hypocalcemia (Metabolism and nutrition disorders) | 22
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22
Diarrhea (Gastrointestinal disorders) | 20
Abdominal pain (Gastrointestinal disorders) | 19
Hypokalemia (Metabolism and nutrition disorders) | 19
Fatigue (General disorders) | 18
Gastroesophageal reflux disease (Gastrointestinal disorders) | 17
Fever (General disorders) | 17
Alopecia (Skin and subcutaneous tissue disorders) | 17
Hypophosphatemia (Metabolism and nutrition disorders) | 16
Back pain (Musculoskeletal and connective tissue disorders) | 16
Peripheral sensory neuropathy (Nervous system disorders) | 14
Insomnia (Psychiatric disorders) | 14
Hyperkalemia (Metabolism and nutrition disorders) | 13
Pain (General disorders) | 12
Dry skin (Skin and subcutaneous tissue disorders) | 12
Upper respiratory infection (Infections and infestations) | 11
Anxiety (Psychiatric disorders) | 11
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11
Sore throat (Respiratory, thoracic and mediastinal disorders) | 11
Hypermagnesemia (Metabolism and nutrition disorders) | 10
Paresthesia (Nervous system disorders) | 10
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 10
Pruritus (Skin and subcutaneous tissue disorders) | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Depression (Psychiatric disorders) | 9
Infusion related reaction (Injury, poisoning and procedural complications) | 8
Non-cardiac chest pain (General disorders) | 8
Weight loss (Investigations) | 8
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8
Oral pain (Gastrointestinal disorders) | 7
Hypercalcemia (Metabolism and nutrition disorders) | 7
Hypoglycemia (Metabolism and nutrition disorders) | 7
Dizziness (Nervous system disorders) | 7
Rash acneiform (Skin and subcutaneous tissue disorders) | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Blurred vision (Eye disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 6
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 6
Sinus tachycardia (Cardiac disorders) | 5
Dental caries (Gastrointestinal disorders) | 5
Edema limbs (General disorders) | 5
Infections and infestations - Other, specify (Infections and infestations) | 5
Mucosal infection (Infections and infestations) | 5
Skin infection (Infections and infestations) | 5
Fall (Injury, poisoning and procedural complications) | 5
Vascular access complication (Injury, poisoning and procedural complications) | 5
Dry eye (Eye disorders) | 4
Colitis (Gastrointestinal disorders) | 4
Esophageal pain (Gastrointestinal disorders) | 4
Malaise (General disorders) | 4
Catheter related infection (Infections and infestations) | 4
Fracture (Injury, poisoning and procedural complications) | 4
Chest wall pain (Musculoskeletal and connective tissue disorders) | 4
Tremor (Nervous system disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 4
Hot flashes (Vascular disorders) | 4
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 4
Thromboembolic event (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MSA states Site is unable to publish until all completed case report forms have been delivered to Sponsor, (Study Completion). Site shall have the right to publish after publication of a multi-center publication coordinated by the Sponsor or (12) mths. after Study Completion; provided, that prior to any such publication or public release of such data, Site shall furnish Sponsor with a copy of any proposed publication at least (45)days in advance of the proposed publication or presentation date.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT01920932/Prot_SAP_002.pdf